CLINICAL TRIAL: NCT01441843
Title: Resistance Under the Microscope; a Randomized Placebo Controlled Parallel Group Design
Brief Title: Resistance Under the Microscope
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Markus Klimek, Vice-head of Anesthesiology, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL3253507810
Record Dates: First submitted 2011-09-22; First posted 2011-09-28 (Estimated); Results first posted 2014-03-10 (Estimated); Last update posted 2023-09-25 (Actual); Status verified 2018-02

CONDITIONS: Anxiety
Keywords: quality of life; lorazepam; anxiety; premedication; surgery; Adult patients; Ambulatory Surgical Procedures; Postoperative Period
MeSH Terms: conditions — Anxiety Disorders | interventions — Lorazepam; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lorazepam (Active Comparator): Lorazepam 4mg/4ml
  Interventions: Drug: Lorazepam
- NaCl 0.9% (Placebo Comparator): NaCl 0.9% 4ml
  Interventions: Drug: NaCl 0.9% (Sodium Chloride)

INTERVENTIONS:
Drug: Lorazepam — Once 1mg <75kg body weight, 1.5mg 75kg and >75kg body weight, IV, before surgery
  Other Names: Temesta
  Arms: Lorazepam
Drug: NaCl 0.9% (Sodium Chloride) — Once 1ml <75kg body weight, 1.5ml 75kg or >75kg body weight, IV, before surgery
  Other Names: NaCl 0.9%
  Arms: NaCl 0.9%

SUMMARY:
The purpose of this study is to determine whether lorazepam, which is used to lower preoperative anxiety, also improves postoperative recovery.

This study data will also be used for further research aiming to identify vulnerable patients in the day-case surgery setting.

DETAILED DESCRIPTION:
Since the early 1980s, the investigators have seen a shift towards day-case surgery. Before surgery, many patients have negative feelings about the surgical procedure. These anxieties have various negative effects. To reduce this resistance preoperative administration of an anxiolytic drug is administered, typically a benzodiazepine. The investigators know that benzodiazepines are effective in reducing anxiety, but up to now there is nog good scientific evidence about the effectiveness of lorazepam on the quality of recovery in day-case surgery patients.

The ultimate goal of our research project is to identify patients who would benefit from preoperative benzodiazepine administration and who not. Identification would substantially contribute to optimal medical decision making.

ELIGIBILITY:
Inclusion Criteria:

* patients > 18 years admitted to the Day-Case Surgery Department Erasmus MC

Exclusion Criteria:

* insufficient command of the Dutch language
* ophthalmology surgery
* Extracorporeal Shock Wave Lithotripsy (ESWL)-, Gastrointestinal endoscopic intervention, Botox-, Abortion and Pain treatment
* Use of psychopharmaceuticals
* Contra-indication of lorazepam use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2010-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Klimek, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus University Medical Center, Rotterdam, Netherlands

REFERENCES:
- [Result] Mijderwijk H, van Beek S, Klimek M, Duivenvoorden HJ, Grune F, Stolker RJ. Lorazepam does not improve the quality of recovery in day-case surgery patients: a randomised placebo-controlled clinical trial. Eur J Anaesthesiol. 2013 Dec;30(12):743-51. doi: 10.1097/EJA.0b013e328361d395. PMID 23635914
- [Derived] Mijderwijk H, Stolker RJ, Duivenvoorden HJ, Klimek M, Steyerberg EW. Clinical prediction model to identify vulnerable patients in ambulatory surgery: towards optimal medical decision-making. Can J Anaesth. 2016 Sep;63(9):1022-32. doi: 10.1007/s12630-016-0673-3. Epub 2016 Jun 9. PMID 27282374

RESULTS

PARTICIPANT FLOW:
Groups:
- Lorazepam: Lorazepam 4mg/4ml
  Lorazepam : Once 1mg <75kg body weight, 1.5mg 75kg and >75kg body weight, IV, before surgery
- NaCl 0.9%: NaCl 0.9% 4ml
  NaCl 0.9% (Sodium Chloride) : Once 1ml <75kg body weight, 1.5ml 75kg or >75kg body weight, IV, before surgery
Period: Overall Study
Arm/Group | Lorazepam | NaCl 0.9%
Started | 200 | 200
Completed | 188 | 195
Not Completed | 12 | 5

BASELINE CHARACTERISTICS:
Population: In retrospect, two patients in the lorazepam group should not have been included due to an administrative error. Data for these two patients were, therefore, excluded from analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lorazepam | NaCl 0.9% | Total
Number analyzed (Participants) | 198 | 200 | 398
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 190 | 191 | 381
  >=65 years | 8 | 9 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (13.7) | 39.3 (13.6) | 39.4 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 85 | 174
  Male | 109 | 115 | 224
Region of Enrollment [Number; unit: participants]
  Netherlands | 198 | 200 | 398

OUTCOME MEASURES:

1. Primary Outcome: Quality of Recovery Score
Description: The Quality of Recovery Score - 40 (QoR-40), a 40-item scale, is used to assess the quality of recovery.
  Each item is rated on a five-point Likert scale (1-5), and the QoR-40 score is calculated as the sum of the scores on these items. Minimal possible score = 40, maximal possible score = 200. A higher score indicates a higher level of quality of recovery.
Time Frame: Baseline; first postoperative working day; seventh postoperative day.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lorazepam | NaCl 0.9%
Number analyzed (Participants) | 188 | 195
scores on a scale
  Seventh postoperative day | 172.8 (21.0) | 176.3 (18.8)
  First postoperative working day | 174.5 (13.0) | 176.4 (12.6)
  Baseline | 177.2 (17.4) | 180.4 (17.5)

2. Secondary Outcome: Anxiety
Description: The State-Trait Anxiety Inventory (STAI) is used to assess anxiety. Scores are calculated by summing the scores on the items, and a higher score indicates a higher level of anxiety.
Time Frame: baseline; after surgery but before discharge; 1 week after surgery
Reporting Status: Not Posted

3. Secondary Outcome: Fatigue
Description: The Multidimensional Fatigue Inventory (MFI) is used to assess the change in fatigue. The MFI is a self-report instrument designed to measure fatigue. Scores are calculated by summing the scores on the items, and a higher score indicates a higher level of fatigue.
Time Frame: baseline; 1 week after surgery
Reporting Status: Not Posted

4. Secondary Outcome: Aggression Regulation
Description: The State-Trait Anger Scale (STAS) is used to assess the aggression regulation. STAS is one of the most used tools for measuring aggression. Scores are calculated by summing the scores on the items, and a higher score indicates a higher level of aggression
Time Frame: baseline; 1 week after surgery
Reporting Status: Not Posted

5. Secondary Outcome: Depressive Mood
Description: The Hospital Anxiety and Depression Scale (HADS) is used to assess the change in depression. The HADS is a well known international outcome measurement for anxiety and depression. It is often used in the clinical setting. Scores are calculated by summing the scores on the items, and a higher score indicates a higher level of depression.
Time Frame: baseline; 1 week after surgery
Reporting Status: Not Posted

6. Secondary Outcome: Somatic Symptoms and Complaints
Description: Medical records are used to assess somatic symptoms and complaints. Next to the medical records, dimensions of the QoR-40 (physical comfort, physical independence and pain) are used to measure somatic symptoms and complaints.
Time Frame: Baseline; first postoperative working day; 1 week after surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Lorazepam | NaCl 0.9%
Serious Adverse Events (participants affected / at risk) | 0/200 | 0/200
Other Adverse Events (participants affected / at risk) | 0/200 | 0/200

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes